CLINICAL TRIAL: NCT07265024
Title: Randomized Controlled Trial on the Effects of Traditional Exercise Programs on the Physical and Mental Health of Visually Impaired Individuals
Brief Title: Traditional Exercise RCT in Visually Impaired Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Normal University (Other)
Collaborators: Changchun University (Unknown)
Responsible Party: Principal Investigator, Guang Yang, Prof. Dr., Prof, Northeast Normal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCEE2026
Record Dates: First submitted 2025-11-20; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Visual Impairments
Keywords: visual impairments; traditional exercise
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Taichi (Experimental)
  Interventions: Behavioral: Baduanjin
- Baduanjin (Experimental)
  Interventions: Behavioral: Taichi
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Taichi — Participants in the Tai Chi group will receive a 12-week simplified 21-form Tai Chi training program. The intervention will consist of supervised sessions conducted three times per week, each lasting approximately 60 minutes. Sessions will include a standardized warm-up, instruction and practice of the 21-form Tai Chi routine, and a brief cool-down period. All training will be delivered by certified Tai Chi instructors experienced in working with individuals with visual impairments. Attendance and adherence will be monitored throughout the intervention period.
  Arms: Baduanjin
Behavioral: Baduanjin — Participants in the Baduanjin group will undergo a 12-week standardized Baduanjin training program. The intervention will be delivered three times per week, with each supervised session lasting approximately 60 minutes. Training sessions will include a structured warm-up, guided practice of the standardized Baduanjin routine, and a brief cool-down period. All sessions will be led by qualified instructors with experience working with visually impaired individuals. Participant attendance and adherence will be recorded throughout the intervention period.
  Arms: Taichi

SUMMARY:
This study aims to investigate the benefits and underlying mechanisms of traditional exercise interventions on the physical and mental health of individuals with visual impairments. A randomized controlled trial design will be employed, enrolling 90 visually impaired participants who will be randomly assigned to one of three groups: a Tai Chi intervention group, a Baduanjin intervention group, or a control group. The Tai Chi group will undergo a 12-week simplified 21-form Tai Chi training program, while the Baduanjin group will receive standardized Baduanjin training. The control group will participate in regular school physical education classes. Eligible participants are university students with visual impairments, defined as having visual acuity ≤ 0.05 or a visual field radius ≤ 10 degrees.

ELIGIBILITY:
Inclusion Criteria:

* University students with visual impairment, defined as visual acuity ≤ 0.05 or a visual field radius ≤ 10 degrees.
* Able to ambulate independently without assistance.
* No severe cardiovascular diseases.

Exclusion Criteria:

* Presence of severe physical illnesses or comorbid conditions that may affect participation.
* History of psychiatric disorders.
* Participation in other structured exercise training programs within the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-01-24 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Single-Leg Stance Test | Month 3
  Assessment of static balance ability by measuring the duration participants can maintain a single-leg stance before and after the intervention.
Timed Up-and-Go (TUG) Test | Month 3
  Evaluation of dynamic balance and functional mobility using the timed up-and-go test, recorded at baseline and post-intervention.
Berg Balance Scale (BBS) | Month 3
  Measurement of overall balance performance using the 14-item Berg Balance Scale, administered before and after the intervention.
Six-Minute Walk Test (6MWT) | Month 3
  Assessment of cardiorespiratory endurance using the six-minute walk test at baseline and following the intervention.
Handgrip Strength Test | Month 3
  Evaluation of upper-limb muscular strength using a calibrated handgrip dynamometer, performed before and after the intervention.
Flexibility Test | Month 3
  Measurement of lower-body flexibility using a standardized sit-and-reach test conducted at baseline and post-intervention.
Self-Rated Depression Scale (SDS) | Month 3
  Assessment of depressive symptoms using the Self-Rated Depression Scale before and after the intervention.
Self-Rated Anxiety Scale (SAS) | Month 3
  Evaluation of anxiety symptoms using the Self-Rated Anxiety Scale administered at baseline and post-intervention.
General Self-Efficacy Scale (GSES) | Month 3
  Measurement of perceived self-efficacy using the General Self-Efficacy Scale at baseline and after the intervention.
WHO Quality of Life-BREF (WHOQOL-BREF) | Month 3
  Assessment of overall quality of life across physical, psychological, social, and environmental domains using the WHOQOL-BREF questionnaire, conducted before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports Science, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided